CLINICAL TRIAL: NCT05672056
Title: Demonstrator in Oral and Maxillofacial Surgery Department
Brief Title: Novel Application of a Low-cost Alternative to Patient Specific Implants (PSI) in Mandibular Free Fibula Flap Reconstruction by Reverse Engineering of Stock Plates: A Pilot Validation Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Ghorab, Demonstrator in Oral and Maxillofacial surgery department, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MohamedGhorabPHD
Record Dates: First submitted 2022-12-30; First posted 2023-01-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Fibula / Surgery; Surgical Flaps; Computer-Aided Design; Mandibular Reconstruction* / Methods; Surgery, Computer-Assisted

STUDY DESIGN:
Intervention Model Description: Pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The intervention will be modifying stock reconstruction plates to mimic patient specific plates in mandibular reconstruction with free fibula flaps
  Interventions: Procedure: Computer guided placement of a stock plate pre-bent on a 3D printed model

INTERVENTIONS:
Procedure: Computer guided placement of a stock plate pre-bent on a 3D printed model — We aim to design a novel guide that can secure the construct of the fibular segments and pre bent plate onto the native mandible and effectively and efficiently translate the VSP into the surgical field.

SUMMARY:
Stock reconstruction plates have been used for decades and represent a tried-and-true alternative to custom plating. Stock plates are readily available, are cost effective, and can be accurately bent before surgery, particularly when using stereolithographic models. Unfortunately, the use of stock plates typically precludes the utilization of predictive holes; this can make inset more difficult as the plates do not precisely match the native mandibular contour. Previous descriptions of fabricating predictive holes with stock plates have been inaccurate and inefficient.

We aim with conducting this research to improve on the ability of pre-bent stock plates of reproducing the VSP in the operating theater allowing accurate native mandible fixation, accurate fibular segments harvest and accurate inset of the reconstruction in lieu of using the expensive alternative of PSI, thus expanding the use of VSP in mandibular reconstruction in resource limited institutions.

DETAILED DESCRIPTION:
Aim of the study:

The aim of the study is to evaluate the accuracy of mandibular reconstruction with free fibula flaps utilizing a novel design of resection and cutting guides based on reverse engineering stock plates into the VSP workflow.

Hypothesis:

The null hypothesis is that there is no significant difference between the postoperatively reconstructed mandible with free fibula flap and the virtually reconstructed mandible preoperatively

PICO:

Population (P): Patients with mandibular segmental defects who will receive free fibula flaps Intervention (I): Three-dimensionally printed guides based on VSP and reverse engineering for resection, predrilling of fixation holes, and shaping of the fibula segments Outcome (O): Accuracy of postoperative mandibular and fibular positions compared with the preoperative virtual surgical plan. In addition to patient reported satisfaction of functional and esthetic outcome. Finally, operative time will be recorded

Trial design:

validity study (pilot study)

Methods A) Participants, interventions & outcomes

Study settings:

The patients will be recruited from the clinics of, the oral and maxillofacial surgery, Cairo University and the Head and neck unit in the National Cancer Institute.

Eligibility criteria:

Inclusion criteria

* Patient with segmental mandibular defects who are planned for free fibula flap reconstruction
* Patients presenting either for immediate reconstruction following resection of tumor or presenting for secondary reconstruction

Exclusion criteria:

* Known allergies or sensitivities to materials such as titanium or acrylic or resin.
* Inability to return for follow up visits.

Post-operative accuracy evaluation:

* Post operative CT scans will be obtained within the first post operative month.
* The post operative DICOM will be segmented in software and the previously designed VSP model will be imported into the project and aligned by best fit algorithm to the unaffected portions of the skull.
* A color heat overlay map will be presented to evaluate the accuracy of reconstruction.

Several anatomical landmarks will be selected to calculate linear deviation measurements.

-Data collection methods Plans for assessment and collection of outcomes will be within the first post operative month and will be done by two assessors independently and inter-examiner calibration will be calculated through Kappa scoring as well as any differences will be solved by consensus. Data management Data will be recorded on diagnostic chart for each patient separately and will be stored with follow up photographs and clinical examination as well as patient's questionnaire. All data will be stored on laptop of the investigator, secured with a password with a backup on google drive and hard copy. The supervisors will have access on the data when needed. Statistical methods Data will be analyzed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 24 (SPSS Inc., Chicago, IL). Numerical data will be described as mean and standard deviation or median and range. Categorical data will be described as numbers and percentages. Chi square test will be used for categorical data. Data will be explored for normality using Kolmogorov-Smirnov test and Shapiro-Wilk test. Comparisons between two groups for normally distributed numeric variables will be done using the paired t-test while for non-normally distributed numeric variables will be done by wilcoxon signed rank test. A p-value less than or equal to 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patient with segmental mandibular defects who are planned for free fibula flap reconstruction
* Patients presenting either for immediate reconstruction following resection of tumor or presenting for secondary reconstruction

Exclusion Criteria:

* Known allergies or sensitivities to materials such as titanium or acrylic or resin.
* Inability to return for follow up visits.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Linear deviation of anatomical landmarks between postoperative outcome and preoperative virtual plan | immediately on the post op CT scans
  Continuous numerical (mm)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University - Faculty of Oral and Dental Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ciocca L, Mazzoni S, Fantini M, Persiani F, Baldissara P, Marchetti C, Scotti R. A CAD/CAM-prototyped anatomical condylar prosthesis connected to a custom-made bone plate to support a fibula free flap. Med Biol Eng Comput. 2012 Jul;50(7):743-9. doi: 10.1007/s11517-012-0898-4. Epub 2012 Mar 24. PMID 22447348
- [Background] Khatib B, Couey M, Patel A, Cheng A, Bell RB. "Custom" Plate in a Day-Accurate Predictive Hole Fabrication Using Point-of-Care 3-Dimensional Printing. J Oral Maxillofac Surg. 2022 Mar;80(3):559-568. doi: 10.1016/j.joms.2021.11.020. Epub 2021 Dec 4. PMID 34958739
- [Background] Mascha F, Winter K, Pietzka S, Heufelder M, Schramm A, Wilde F. Accuracy of computer-assisted mandibular reconstructions using patient-specific implants in combination with CAD/CAM fabricated transfer keys. J Craniomaxillofac Surg. 2017 Nov;45(11):1884-1897. doi: 10.1016/j.jcms.2017.08.028. Epub 2017 Sep 5. PMID 28965991